CLINICAL TRIAL: NCT01999569
Title: The Role of Estrogen in Luteinizing Hormone Surge and Ovulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: LH-2013
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-10

CONDITIONS: Ovulation Disorder; Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts | interventions — Letrozole

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control cycle. No intervention.
- Letrozole (Experimental): 5mg daily
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole administered daily through the time of ovulation.
  Other Names: Femara
  Arms: Letrozole

SUMMARY:
The purpose of the study is to establish that sustained estrogen levels are the driving force for the LH surge, and are thereby necessary for ovulation to occur. We predict that by reducing levels of circulating estrogen, letrozole, an aromatase inhibitor, will inhibit ovulation from occurring.

DETAILED DESCRIPTION:
Sine the common understanding of ovulation in a natural cycle suggests that a sustained, elevated estradiol level is required to trigger the LH surge, administration of letrozole throughout the cycle should lower estradiol levels and prevent the LH surge from occurring. In this study, we sought to determine if the LH surge, ovulation and luteinization occurs in spite of low estradiol levels by daily administration of letrozole in a group of normal ovulatory volunteers in a prospective study.

After IRB approval and informed consent were obtained, ten willing volunteers that met inclusion criteria (no hormonal contraception within 3 months, regular menstrual cycles 26 - 30 days, normal thyroid function and normal prolactin, and no pregnancy currently or within 3 months) were monitored for one month without treatment for evaluation of normal ovulation.

Natural control cycle The subjects used home urine LH tests (Clearblue® Easy, SPD Swiss Precision Diagnostics, Switzerland) on days 10-18 to monitor for the LH surge in both the initial natural cycle and the letrozole cycle. Blood was drawn every other day starting on day 12 of the cycle through day 22 to measure estradiol and progesterone levels, and follicular development was monitored using transvaginal ultrasound on cycle day 12-14.

Letrozole cycle In the next cycle, all ten subjects were administered oral letrozole 5 mg daily (Femara®, Novartis Pharmaceuticals Corporation, East Hanover, NJ ) starting on cycle day 1-3 and continuing through the completion of the study (cycle day 22). Once again, serum estradiol and progesterone levels were measured every other day on days 12-22. The development of the ovarian follicles was monitored by transvaginal ultrasound once in each cycle between days 12-14, and LH surge was monitored with home urine ovulation tests on days 10-18. Table 1 illustrates protocols for both the natural control cycle and the letrozole study cycle.

The primary outcome, assessment of ovulation in letrozole cycles, was determined by the presence or absence of progesterone elevation (>1.5 ng/mL) and the presence or absence of a positive urinary LH test. The bioequivalence evaluation of two cycles (before and after letrozole administration) was based on pharmacokinetic parameters such as area under the serum concentration-time curve (AUC), the peak serum concentration (Cmax) and the time of peak serum concentration (Tmax). Cmax and Tmax were determined by visual inspection from each volunteer's serum concentration-time curve for estradiol and progesterone. AUC was calculated by the linear trapezoidal method from day 12 through day 22 in both the initial natural cycle and the letrozole cycle.

Paired t-tests, or Wilcoxon Signed Rank tests if non-normally distributed, were used to evaluate the statistical significance of the mean values of the pharmacokinetic parameters. The McNemar test was used to assess the difference in LH surge and follicular development before and after letrozole administration. A standard of statistical significance (alpha) of 0.05 was used in all cases. The SAS System (SAS Institute, Cary, NC) was used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient having regular menstrual cycles between 26-30 days
* Ages 18-40
* Patient must not be sexually active during the study period, or if so must be using a reliable form of non-hormonal birth control including tubal ligation or vasectomy, non-hormonal intrauterine contraceptive device (IUD), or condoms with spermicide.
* Willing to participate in study and available for all monitoring visits.
* IRB consent

Exclusion Criteria:

* Patient must NOT have used hormonal contraception three months or less prior to study.
* Irregular menstrual cycles (<26 days or >30 days within the last 6 months.
* Untreated thyroid dysfunction or hyperprolactinemia
* Pregnancy (current or within 3 months) or breastfeeding
* Allergy or contraindication to letrozole

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Hurst, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Women's Institute at Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen A, Bentley GE, Cabrera R, Ortega HH, Perfito N, Wu TJ, Micevych P. Hormonal regulation of female reproduction. Horm Metab Res. 2012 Jul;44(8):587-91. doi: 10.1055/s-0032-1306301. Epub 2012 Mar 21. PMID 22438212
- [Background] Morioka N, Zhu C, Brannstrom M, Woessner JF, LeMaire WJ. Mechanism of mammalian ovulation. Prog Clin Biol Res. 1989;294:65-85. PMID 2657783
- [Background] Goh HH, Ratnam SS. The LH surge in humans: its mechanism and sex difference. Gynecol Endocrinol. 1988 Jun;2(2):165-82. doi: 10.3109/09513598809023624. PMID 3055821
- [Background] Laven JS, Fauser BC. What role of estrogens in ovarian stimulation. Maturitas. 2006 Jul 20;54(4):356-62. doi: 10.1016/j.maturitas.2006.04.022. Epub 2006 Jun 19. PMID 16782289
- [Background] Casper RF, Mitwally MF. Review: aromatase inhibitors for ovulation induction. J Clin Endocrinol Metab. 2006 Mar;91(3):760-71. doi: 10.1210/jc.2005-1923. Epub 2005 Dec 29. PMID 16384846
- [Background] Mitwally MF, Casper RF. Aromatase inhibition reduces the dose of gonadotropin required for controlled ovarian hyperstimulation. J Soc Gynecol Investig. 2004 Sep;11(6):406-15. doi: 10.1016/j.jsgi.2004.03.006. PMID 15350255
- [Background] Burstein HJ, Griggs JJ, Prestrud AA, Temin S. American society of clinical oncology clinical practice guideline update on adjuvant endocrine therapy for women with hormone receptor-positive breast cancer. J Oncol Pract. 2010 Sep;6(5):243-6. doi: 10.1200/JOP.000082. Epub 2010 Aug 6. PMID 21197188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ovulatory volunteers
Groups:
- Control Then Letrozole: Control cycle. Then letrozole cycle
Period: Control Cycle
Arm/Group | Control Then Letrozole
Started | 10 (First cycle no meds)
Completed | 10
Not Completed | 0
Period: Letrozole Treatment Cycle
Arm/Group | Control Then Letrozole
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Control cycle. Then letrozole cycle
Arm/Group | Control
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progesterone Level Greater Than 1.5 ng/mL
Description: Serum progesterone ng/mL drawn during cycle days twelve through 22
Time Frame: Cycle days 12-22
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control cycle
Arm/Group | Control | Letrozole Treatment Cycle
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

2. Secondary Outcome: Number of Participants With a Positive LH Test
Description: Urine ovulation tests assessed
Time Frame: Cycle days 10-18
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Letrozole Treatment Cycle
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

3. Secondary Outcome: Number of Participants With Follicular Development
Description: Ovulation; elevated progesterone
Time Frame: Cycle day 12
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Letrozole Treatment Cycle
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: two ovulation cycles (2 months)
Arm/Group | Control | Letrozole
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No